CLINICAL TRIAL: NCT02705703
Title: Phase I/II Study of Low-Dose Cyclophosphamide, Tumor Associated Peptide Antigen (TAPA)-Pulsed Dendritic Cell (DC) Therapy and Low Dose GM-CSF, as Consolidation Therapy in Patients With Metastatic Solid Malignancies
Brief Title: Consolidation Therapy in Patients With Metastatic Solid Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue study.
Sponsor: Kiromic BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KiroVAX004; BSK01 Dendritic cell vaccine (Other: Kiromic)
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Metastatic Solid Malignancies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAPA-pulsed DC vaccine (Experimental): The subject will take low-dose cyclophosphamide by mouth for 5 days starting 7 days prior to the vaccine cycle. The vaccine contains 1 x 10^7 TAPA-pulsed dendritic cells and is administered SQ with low-dose GM-CSF following the low-dose cyclophosphamide cycle. A total of six (6) cycles of cyclophosphamide and six (6) DC vaccines cycles will be administered alternating every 14 days.
  Interventions: Biological: TAPA-pulsed DC vaccine

INTERVENTIONS:
Biological: TAPA-pulsed DC vaccine — A cycle of low-dose cyclophosphamide (100mg/day) by mouth for 5 days starting seven 7 days prior to the DC vaccine cycle to reduce Treg activity. Low-dose cyclophosphamide will be taken every 14 days for six 6 cycles. A total of 6 vaccines containing 1 x 10^7 TAPA-pulsed DC will be administered SQ every 14 days. The DC vaccine is given on Day 1 of the DCV cycle plus low-dose GM-CSF 50mcg/day SQ x 5 days (Day 1 to Day 4). GM-CSF is administered for 5 days to increase monocyte production and dendritic cell precursors to optimize immune responses.

SUMMARY:
This study evaluates the effectiveness of Tumor Associated Peptide Antigens (TAPA) pulsed dendritic cell injections as a potential consolidation therapy for patients with metastatic solid malignancies (SM). The investigators hypothesize that treatment of patients with metastatic SM who demonstrate a tumor response, or whose disease remains stable, after conventional first-line systemic therapy AND who lack an available, potentially curative therapeutic intervention and whose tumor cells and/or blood express at least one (1) TAPA of a defined panel of TAPAs will result in TAPA-specific T-cell responses without significant toxicities. The investigators also hypothesize CD4+ and CD8+ T-cell responses generated against specific TAPAs may translate into clinical antitumor activity.

DETAILED DESCRIPTION:
Patients diagnosed with metastatic solid malignancies (SM), who have responded or whose disease remains stable following first line systemic therapy, and without available, potential curative therapeutic options, will be candidates for this Phase I/II study. Potentially eligible patients who agree to participate and sign a consent form will have their neoplastic cells and/or blood analyzed for the expression of a specific panel of Tumor Associated Peptide Antigens (TAPAs), including Sp17, ropporin, AKAP-4, PTTG1, Span-xb, Her-2/neu, HM1.24, NY-ESO-1 and MAGE-1. Patients whose tumors express one (1) or more of these TAPAs will receive three (3) days of subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) to increase bone marrow production of monocytes and dendritic cell (DC) precursors, and whole blood will be obtained by phlebotomy and/or leukapheresis for generation of autologous DCs. Patient's DCs will be generated in Kiromic's Cell Processing Good Manufacturing Process (GMP) facility, according to established Standard Operating Procedures, and activated by pulsing/loading them with the TAPA(s) relevant for each particular patient. Patients will receive five (5) days of low-dose cyclophosphamide prior to each vaccination with TAPA-pulsed DCs to decrease Treg activity. TAPA-pulsed DCs will be administered at a fixed dose of up to 1 X 107 DCs at least two (2) days following cyclophosphamide administration. DC vaccination schedule will be once every fourteen (14) days via subcutaneous (SC) and intradermal (ID) injections for a total of 6 vaccinations. Low dose GM-CSF will also be administered SC for five (5) consecutive days, starting three (3) to six (6) hours after each TAPA-pulsed DC treatment, to optimize immune responses. Patients will be followed on a weekly basis (or more frequently if required) to evaluate treatment-related toxicity. Immune responses and anti-tumor responses will be evaluated per protocol specifications. Continuation and stopping rules for the study will be defined based on toxicity/tolerability (Phase I) and/or immune responses (Phase II).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Patients at least eighteen (18) years of age with histologically proven metastatic solid malignancies (SM) AND whose SM demonstrates a response, or whose disease remains stable, after conventional, first-line systemic therapy, AND who lack any available, potentially curative therapeutic intervention, will be eligible for participation in this study.
3. Expression of one (1) or more of the following TAPAs; Sp17, AKAP-4, Ropporin, PTTG-1, Span-xb, Her-2/neu, HM1.24, NY-ESO-1 and MAGE-1, by either reverse transcriptase polymerase chain reaction (RT-PCR) and/or immunocytochemistry, Western blotting or ELISA, in neoplastic cells and/or blood. For HER-2/neu expression, positive FISH results are acceptable. All lab tests will be performed in a CLIA certified facility
4. Presence of measurable or evaluable disease.
5. Patients must not have any active infectious process.
6. Patients must have a negative test for HIV, Hepatitis A, B, and C.
7. Patients must not be receiving active immunosuppressive therapy.
8. Patients must have discontinued systemic antineoplastic therapy (including endocrine and biological agents, as well as systemic corticosteroids) at least three (3) to four (4) weeks prior to enrollment. Toxicities from previous therapies must be grade 1 or less.
9. Patients may not have any known allergy to GM-CSF.
10. Patients must be willing to provide at least 250 mls of whole blood obtained by phlebotomy and/or consent to leukapheresis for DC generation.
11. Adequate renal and hepatic function (creatinine ≤ 2.0 mg/dl, bilirubin ≤ 2.0 mg/dl, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 4X upper limit of normal range).
12. Adequate hematologic function (Platelets ≥ 60,000/mm3, lymphocytes ≥ 1,000 mm3, neutrophils ≥ 750/mm3, hemoglobin ≥ 10.0 g/dl).
13. Karnofsky performance status ≥ 70%.
14. Expected survival ≥ 6 months.
15. Patient Human Leucocyte Antigen (HLA) typing should demonstrate HLA-A*01, and/or HLA-A*02, and/or HLA-A*24 subtype restriction.
16. Either a female or male of reproductive capacity wishing to participate in this study must be using, or agree to use, one or more types of birth control during the entire study and for 3 months after completing the study. Birth control methods may include condoms, diaphragms, birth control pills, spermicidal gels or foams, anti-gonadotropin injections, intrauterine devices (IUD), surgical sterilization, or subcutaneous implants. Another choice is for a subject's sexual partner to use one of these birth control methods. Women of reproductive capacity will be required to undergo a urine pregnancy test before completion of the post-screening informed consent process.

Exclusion Criteria:

1. Patients without confirmed metastatic SM and/or response to conventional, first-line systemic therapy using standard RECIST criteria, or patients with confirmed metastatic SM and/or response to conventional, first-line systemic therapy using standard RECIST criteria, but who have an available, potentially curative therapeutic option will be excluded from participation in this study.
2. Patients without measurable or evaluable disease.
3. Patients receiving cytotoxic therapy (including endocrine and biological agents), radiation therapy, immunotherapy or non-topical steroids, within three (3) weeks of enrollment.
4. Active immunosuppressive therapy (excluding topical steroids) for any other condition.
5. Persistent fever (>24 hours) documented by repeated measurement or active, uncontrolled infection within 4 weeks of enrollment.
6. Active ischemic heart disease or history of myocardial infarction within six months.
7. Active autoimmune disease, including, but not limited to, Systemic Lupus Erythematosus (SLE), Multiple Sclerosis (MS), Ankylosing Spondylitis (AS), and Rheumatoid Arthritis (RA).
8. Pregnancy or breast feeding.
9. Active second invasive malignancy, other than basal cell carcinoma of the skin.
10. Life expectancy ≤ 6 months.
11. Patients with contraindications to CYP and/or GM-CSF.
12. History of allergy to CYP and/or GM-CSF.
13. Patients who have received organ transplants.
14. Patients with psychological or geographic conditions that prevent adequate follow-up or compliance with the study protocol.
15. Patients diagnosed with central nervous system (CNS) metastases or involvement at any time during disease course are excluded from the study.
16. Patient with HLA alleles not belonging to any of the following subtypes: HLA-A*01, or HLA-A*02, or HLA-A*24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events due to administration of TAPA-pulse DC vaccine | every 7 days up to 5 months

SECONDARY OUTCOMES:
Immunological efficacy as indicated by T-cell cytokine levels | up to 5 months
Immunological efficacy as determined by a positive delayed type hypersensitivity (DTH) skin test | up to 5 months